CLINICAL TRIAL: NCT04253249
Title: Endoscopic Ultrasound Guided Pancreatic Cyst Ablation With a Monopolar Radiofrequency Ablation Probe
Brief Title: Pancreatic Cyst Ablation With a Monopolar Radiofrequency Ablation Probe
Status: Withdrawn | Type: Observational
Why Stopped: No funding was obtained.
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Mohamed Othman, Associate Professor, Baylor College of Medicine
Other Study IDs: H-38304
Record Dates: First submitted 2020-01-27; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Treatment Related Cancer
MeSH Terms: conditions — Neoplasms, Second Primary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pancreatic cysts (A cyst is a thin walled cavity containing fluid) were rarely reported previously, but have been on a rise due to advanced imaging for evaluating pancreatic lesions or other medical reasons has increased detection of pancreatic cysts. Study shows transformation of pancreatic cysts to be 10.8 for every 100,000 women and 13.8 for every 100,000 men.

Pancreatic cysts are divided in two groups; serous and mucinous. Serous cysts are thin walled cysts and are not associated with precancer. On the other hand, mucinous cysts have a tendency to progress to pancreatic cancer.

Radio frequency ablation (RFA) is an alternative method used for patients who could not or decided to not undergo surgical removal of the cyst. This study is a standard of care study and no changes in regards to the procedure scheduled with the physician will be changed.

DETAILED DESCRIPTION:
Pancreatic cysts were rarely reported previously, however, the increased use of advanced imaging techniques (mainly computerized topography and magnetic resonance imaging), for evaluating suspected pancreatic pathology or for other medical reasons has increased the detection of pancreatic cysts. Prevalence can range from 2.5-38% (1,3). These rates vary by patient's age and modality of imaging used (i.e: CT vs MRI). The rate of a malignant transformation in pancreatic cysts is not well known, however, very low. A study using the SEER data reported this rate to be 10.8 for every 100,000 women, or 13.8 for every 100,000 men with more than 85% of malignancies being detected in patient's age 40-84 years of age. (4) The most common histological type was adenocarcinoma, with mucinous producing tumors making about 4% of all adenocarcinomas detected. Pancreatic cysts are categorized under two major groups; serous and mucinous. Serous cystadenomas are thin walled cysts and are not associated with precancer. Mucinous cysts on the other hand have various diameters and contain viscous fluids which have the tendency to progress to pancreatic cancer. Radiofrequency ablation was recently proposed as an alternative for patients who could not or would not undergo surgical resection. In a recent study under the title "Endoscopic ultrasound guided radiofrequency ablation, for pancreatic cystic neoplasms and neuroendocrine tumors", eight patients with pancreatic cystic lesions were recruited for the study. Six patients had pancreatic cystic neoplasm. Post procedure imaging in 3-6 months showed complete resolutions of the cysts in 2 cases after using EUS RFA. No major complications were observed within 48 hours after the procedure, and two patients had mild abdominal pain which was resolved within 3 days after the surgery. (1) Management of pancreatic cysts includes surgical or non-surgical, or can be observational with repeat imaging. Management type depends on factors including pathologic features of the cyst on imaging (cyst size, enhancing cyst walls, duct size…etc), and the patient's ability to undergo surgery. Older patients with preexisting morbidities may not be eligible for a surgical resection, thus the use of endoscopic ultrasound interventions maybe appropriate. Endoscopic ultrasound guided radio frequency ablation has been used in treating certain pancreatic lesions, with a favorable pancreatic outcome (5)

ELIGIBILITY:
Inclusion Criteria:

-Adult (18-64 yrs), Geriatric (65+ yrs)

Exclusion Criteria:

* Pregnant woman
* Neonates
* Children

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Groups to be recruited will include:
  Patients
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-05-19 (Estimated); Study Completion 2020-12-19 (Estimated)

PRIMARY OUTCOMES:
Treatment pancreatic cyst without surgery | Through study completion, an average of 1 year
  Efficacy of managing pancreatic cyst without open surgery

CONTACTS AND LOCATIONS:
Overall Officials: MOHAMED O. OTHMAN, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided